CLINICAL TRIAL: NCT06474494
Title: Clinical Evaluation of the Effect of Double Layer Application Using a Universal Adhesive in Restorations of Non-carious Cervical Lesions: Double-blind Randomized Clinical Trial
Brief Title: Evaluation of Double Layer Application Using a Universal Adhesive in the Quality of Cervical Lesions Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Principal Investigator, Mario Felipe Gutiérrez Reyes, Associate Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEC2024050
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Non-carious Cervical Lesions
Keywords: Dental bonding; Tooth erosion; Tooth wear; Adhesive systems; Double layer
MeSH Terms: conditions — Tooth Erosion; Tooth Wear

STUDY DESIGN:
Intervention Model Description: This is a four-arm, double-blind, randomized controlled clinical trial. Experimental group 1: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying a double layer of Scotchbond Universal Plus adhesive applied as etch-and-rinse mode.
  Experimental group 2: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying a double layer of Scotchbond Universal Plus adhesive applied as selective enamel etching mode.
  Control group 1: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying one layer of Scotchbond Universal Plus adhesive applied as etch-and-rinse mode.
  Control group 2: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying one layer of Scotchbond Universal Plus adhesive applied as selective enamel etching mode.
  LCNCs will be randomized to application mode and number of layers
Who Masked: Participant, Outcomes Assessor
Masking Description: Two blinded, experienced, and calibrated dentists (who specialized in esthetic dentistry with more than 15 years of clinical practice), will perform the clinical evaluation. Patients will be also blinded to group assignment. An inter-examiner and inter-examiner agreement of at least 85% will be necessary before beginning the evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Experimental group 1 (Experimental): 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying double layer of Scotchbond Universal Plus adhesive applied as etch-and-rinse mode
  Interventions: Procedure: Application of double layer; Procedure: Etch-and-rinse application mode
- Experimental group 2 (Experimental): 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying double layer of Scotchbond Universal Plus adhesive applied as selective enamel etching mode
  Interventions: Procedure: Application of double layer; Procedure: Selective enamel etching application mode
- Control group 1 (Active Comparator): 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying one layer of Scotchbond Universal Plus adhesive applied as etch-and-rinse mode
  Interventions: Procedure: Application of one layer; Procedure: Etch-and-rinse application mode
- Control group 2 (Active Comparator): 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying one layer of Scotchbond Universal Plus adhesive applied as selective enamel etching mode
  Interventions: Procedure: Application of one layer; Procedure: Selective enamel etching application mode

INTERVENTIONS:
Procedure: Application of one layer — 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying one layer of Scotchbond Universal Plus adhesive
  Arms: Control group 1; Control group 2
Procedure: Application of double layer — 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying double layer of Scotchbond Universal Plus adhesive
  Arms: Experimental group 2; Experimental: Experimental group 1
Procedure: Etch-and-rinse application mode — 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying Scotchbond Universal Plus adhesive applied as etch-and-rinse application mode
  Arms: Control group 1; Experimental: Experimental group 1
Procedure: Selective enamel etching application mode — 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying Scotchbond Universal Plus adhesive applied as selective enamel etching mode
  Arms: Control group 2; Experimental group 2

SUMMARY:
The aim of this study will be to evaluate the effect of a double layer application of a universal adhesive system used as etch-and-rinse application mode in non-carious cervical lesions (NCCLs), on the 6- and 12-months clinical performance.

Materials & Methods: 144 restorations were randomly placed in 36 subjects (16 male and 20 female) according to the following groups (n=36): ER1 (one layer of Scotchbond Universal Plus adhesive applied as etch-and-rinse mode); ER2 (double layer of Scotchbond Universal Plus adhesive applied as etch-and-rinse mode); SEE1 (one layer of Scotchbond Universal Plus adhesive applied as selective enamel etching); SEE2 (double layer of Scotchbond Universal Plus adhesive applied as selective enamel etching). All groups were light-cured for 10s/1,000 mW/cm2 only after final layer. A resin composite will be placed by applying three increments and each one will be light cured for 20s/1,000 mW/cm2. The restorations will be finished immediately with fine diamond burs and polishers. The restorations will be evaluated at baseline and after 6- and 12-months by using the FDI criteria. The following outcomes will be evaluated: retention, marginal staining, marginal adaptation, post-operative sensitivity and recurrence of caries. The differences among the groups will be calculated using Friedman repeated measures analysis of variance rank (α = 0.05).

DETAILED DESCRIPTION:
This is a four-arm, double-blind, randomized controlled clinical trial. Experimental group 1: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying a double layer of Scotchbond Universal Plus adhesive applied as etch-and-rinse mode.

Experimental group 2: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying a double layer of Scotchbond Universal Plus adhesive applied as selective enamel etching mode.

Control group 1: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying one layer of Scotchbond Universal Plus adhesive applied as etch-and-rinse mode.

Control group 2: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations applying one layer of Scotchbond Universal Plus adhesive applied as selective enamel etching mode.

LCNCs will be randomized to application mode and number of layers. All groups will be light-cured with a light-curing device (SmartLite Focus, Dentsply) with a light intensity of 900 mW/cm² for 10 seconds. Operators will restore the cervical area by applying three increments of resin (Filtek Supreme XT, 3M). Each increment will light cure for 20 s at 900 mW/cm2 (SmartLite Focus, Dentsply). Restorations will be finished immediately with fine and extra fine diamond burs and polished with polishing spirals.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Presence of at least two Non-Carious Cervical Lesions in the dental arch with a need for restorative treatment.
* Acceptable level of oral hygiene according to the Simplified Oral Hygiene Index.
* At least 20 teeth in function.
* Non-Carious Cervical Lesions with a maximum of 50% of enamel margin.

Exclusion Criteria:

* Driving difficulties that prevent adequate oral hygiene.
* Periodontal disease.
* Active caries lesions on the teeth included in the research.
* Parafunctional habits.
* Active staples of removable partial dentures on the teeth included in the research and that these are not pillars of prostheses.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Retention rate of restorations | From date of randomization until twenty four months
  Retention rate measured by World Dental Federation (FDI) criteria as following:
  * G: Clinically good - Small hairline crack;
  * SS: Clinically sufficient/satisfactory - Two or more or larger hairline cracks and/or chipping (not affecting the marginal integrity);
  * US: Clinically unsatisfactory - Chipping fractures which damage marginal quality; bulk fractures with or without partial loss (less than half of the restoration);
  * PO: Clinically poor - (Partial or complete) loss of restoration, (replacement necessary).

SECONDARY OUTCOMES:
Marginal Adaptation rate of restorations | From date of randomization until twenty four months
  Marginal Adaptation rate measured by World Dental Federation (FDI) criteria as following:
  * VG: Clinically very good - Harmonious outline, no gaps, no discoloration;
  * G: Clinically good - Small marginal fracture removable by polishing;
  * SS: Clinically sufficient/satisfactory - Several small enamel or dentin fractures;
  * US: Clinically unsatisfactory - Notable enamel or dentine wall fracture;
  * PO: Clinically poor - Filling is loose but in situ.
Marginal Staining rate of restorations | From date of randomization until twenty four months]
  Marginal Staining rate measured by World Dental Federation (FDI) criteria as following:
  * VG: Clinically very good - No marginal staining;
  * G: Clinically good - Minor marginal staining, easily removable by polishing;
  * SS: Clinically sufficient/satisfactory - Moderate marginal staining, not esthetically unacceptable;
  * US: Clinically unsatisfactory - Pronounced marginal staining; major intervention necessary for improvement;
  * PO: Clinically poor - Deep marginal staining not accessible for intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mario Felipe Gutierrez Reyes, Study Director — Universidad de los Andes, Chile
Locations (1):
- Mario Felipe Gutiérrez Reyes, Santiago, Santiago Metropolitan, Chile